CLINICAL TRIAL: NCT05016895
Title: The Resiliency Through Azithromycin for Children Project: Implementation Research on Bi-Annual Mass Distribution of Azithromycin to Children 1-11 Months in Côte d'Ivoire
Brief Title: REACH2: Implementation Research on Bi-Annual Mass Distribution of Azithromycin to Children 1-11 Months in Côte d'Ivoire
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Ministry of Health, Ivory Coast (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1743615
Record Dates: First submitted 2021-08-03; First posted 2021-08-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Child Mortality
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bi-annual single dose azithromycin (Experimental): Mass, community-based distribution of single dose azithromycin solution (200 mg/5ml) dosed at 20 mg/kg weight to all eligible infants ages 1 to 11 months twice yearly (approximately 6 months apart)
  Interventions: Drug: Single-dose azithromycin

INTERVENTIONS:
Drug: Single-dose azithromycin — Bi-annual mass, community-based distribution of single-dose azithromycin to children ages 1 to 11 months.

SUMMARY:
REACH2 is a three-year implementation research study designed to examine the implementation through a mass drug administration platform of bi-annual single-dose azithromycin to reduce child mortality among children ages 1 to 11 months who reside in high child mortality settings.

DETAILED DESCRIPTION:
The aim of the study is to provide the government of Côte d'Ivoire and other stakeholders the information needed to understand what is required to bring bi-annual mass drug administration (MDA) of single-dose azithromycin for children ages 1 to 11 months in high child mortality settings to scale using the existing MDA platform used for trachoma and other neglected tropical diseases.

Design: The serial cross-sectional study will be carried out in 19 health districts in coordination with the trachoma MDAs over the course of three years. The intervention under study will involve a public health campaign of bi-annual distribution of single-dose azithromycin, including:

1. Expanded coverage with azithromycin during annual trachoma MDAs to children 1-5 months of age when delivered at the same time as the annual trachoma MDA, which already covers children 6-11 months, followed by
2. Stand-alone MDAs targeting children 1 to 11 months delivered at the approximately 6-month interval between annual trachoma MDAs, or bi-annually in areas where the annual trachoma MDAs are phased out.

To study scale up of these intervention activities, the investigators will systematically collect data, guided by the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) implementation science framework. Data collection activities will involve:

1. Analyses of routine monitoring, process, and adverse drug reaction data from the trachoma MDA platform into which the REACH activities are being integrated
2. Periodic, cross-sectional, post-MDA surveys to verify coverage and examine exposure to project information/messaging
3. Qualitative data collection through in-depth interviews (IDI) and/or focus group discussions (FGD) with parents or primary caregivers of children ages 1 to 11 months in the 19 health districts, and district-level MDA implementers to explore issues of acceptability, communication, challenges and areas for improvement in implementation.

Further, after the first round of the annual trachoma MDA scheduled to take place in July 2021, a round of focus groups will be carried out with parents of children ages 1-11 months and local implementers to inform message development for the public health campaign.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 to 11 months
* Resident in targeted community

Exclusion Criteria:

* Children below 3.0 kg (3rd centile for healthy 1-month old infants in the WHO growth charts)
* Appears seriously ill at the time of the MDA (per the CDD's assessment)
* Unable to swallow liquid delivered through a needle-less syringe because of physical limitations
* Known allergy to macrolides, including azithromycin, based on the primary caregiver's report of prior adverse reaction to medication likely to be a macrolide
* prior allergic reaction to medication likely to be a macrolide

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 767535 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
% of eligible population covered by intervention | three years
  coverage of the intervention's target population (reach) with azithromycin in targeted health districts
Infant mortality rate | three years
  Rate of child deaths among children under 1 year of age per 1,000 population
Implementation fidelity | three years
  Proportion of intervention activities are carried out as planned

SECONDARY OUTCOMES:
Cost of the program as a whole | three years
  Program costs will be calculated based on the following inputs: personnel, supplies/recurrent goods, capital goods, travel/transport, space, services, and training
Cost per child treated | three years
  Program costs per child treated
Cost per death averted | three years
  Program costs per death averted

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dulli, PhD, Principal Investigator — FHI 360
Locations (1):
- FHI 360, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
Quantitative survey data from the study will be shared. These data contain no individually identifying data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be shared indefinitely within 6 months of the conclusion of the study.
Access Criteria: Data will be made publicly available on Harvard Dataverse.